CLINICAL TRIAL: NCT05642559
Title: Retrospective and Prospective Observational Study for the Development and Validation of Chronic Cough Patient Perspective Questionnaire
Brief Title: Study for the Development and Validation of Chronic Cough Patient Perspective Questionnaire
Acronym: MISP
Status: Completed | Type: Observational
Sponsor: Ospedale Policlinico San Martino (Other)
Responsible Party: Principal Investigator, BRAIDO, Professor, Ospedale Policlinico San Martino
Other Study IDs: 22/2022
Record Dates: First submitted 2022-11-10; First posted 2022-12-08 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Chronic Cough
MeSH Terms: conditions — Chronic Cough | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — Assessment of refractory chronic cough (RCC) or unexplained chronic cough (UCC) impact on HRQoL of the explored population and relationship with clinical variables. Development of a web application of the questionnaire.

SUMMARY:
Starting from Chronic Cough Impact Querstionnaire (CCIQ), of which we are the authors and copyright holders, it will be developed and validated a shortened version with psychometric properties allowing the use in the evaluation of single patient (Chronic Cough Patient Perspective).

The CCPP will allow to unmask the problem, reduce underdiagnosis, increase awareness on chronic cough, measure the impact of the chronic cough and its treatments on the patient's life.

ELIGIBILITY:
Inclusion Criteria:

diagnosis of RCC (Residual Cough VAS:>10/100 mm) according to ERS guidelines

Exclusion Criteria:

difficulty in understanding the italian language in both spoken and written form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients (>18 years) suffering from RCC (Residual Cough VAS:>10/100 mm)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Chronic Cough Impact Questionnaire (CCIQ) | february 2023
  To develop the preliminary CCPP questionnaire starting from Chronic Cough Impact Questionnaire (CCIQ) (2) and available database

SECONDARY OUTCOMES:
Chronic Cough Impact Questionnaire (CCIQ) | August 2023
  Assessment of refractory chronic cough (RCC) or unexplained chronic cough impact on HRQoL of the explored population and relationship with clinical variables

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Martino, Genova, Italy